CLINICAL TRIAL: NCT01622348
Title: A Randomized, Double-Blind, Placebo-Controlled, 4-week Trial of IMO-3100 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Trial of IMO-3100 in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3100-202
Record Dates: First submitted 2012-05-21; First posted 2012-06-19 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Actively Extending Plaque Psoriasis; Moderate to Severe Plaque Psoriasis
Keywords: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Saline for Injection
  Interventions: Drug: Saline for Injection
- IMO-3100 at 0.16 mg/kg (Active Comparator): IMO-3100 at 0.16 mg/kg SC once weekly based on body weight at screening, not to exceed 20 mg per injection
  Interventions: Drug: IMO-3100 at 0.16 mg/kg
- IMO-3100 at 0.32 mg/kg (Active Comparator): IMO-3100 at 0.32 mg/kg SC q wk x 4 wk based on body weight at screening, not to exceed 40 mg per injection
  Interventions: Drug: IMO-3100 at 0.32 mg/kg

INTERVENTIONS:
Drug: IMO-3100 at 0.16 mg/kg — IMO-3100 at 0.16 mg/kg SC q wk x 4 wks based on body weight at screening, not to exceed 20 mg per injection
  Arms: IMO-3100 at 0.16 mg/kg
Drug: Saline for Injection — Saline for Injection 0.01 mL/kg SC q wk x 4 wk based on body weight at screening, not to exceed 1.25 mL
  Arms: Placebo
Drug: IMO-3100 at 0.32 mg/kg — IMO-3100 at 0.32 mg/kg SC q wk x 4 wks based on body weight at screening, not to exceed 40 mg per injection
  Arms: IMO-3100 at 0.32 mg/kg

SUMMARY:
The purpose of this study is to evaluate different dose levels of IMO-3100 compared to placebo administered for 4 weeks to patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability and treatment effect of different dose levels of IMO-3100 compared to placebo administered for 4 weeks to patients with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Is age 18 to 70 years, inclusive;
* Completes the informed consent procedure (see Section 15.3), including signing and dating the informed consent form;
* Has moderate to severe plaque psoriasis meeting the criteria specified above;
* Female subjects must have a negative pregnancy test at screening and on Day 1 prior to start of treatment;
* Female subjects of childbearing potential (see Section 8.4.1) and male subjects who have partners of childbearing potential must agree to use effective birth control (contraception; see Section 8.4.1) from Screening through the treatment period and for four (4) weeks after the last injection of study drug.

Exclusion Criteria:

* Has known hypersensitivity to any oligodeoxynucleotide;
* Is nursing;
* Has body weight < 50 kg;
* Has BMI > 34.9 kg/m2;
* Regularly consumes > 3 drinks of alcoholic beverages (beer, wine, or distilled spirits) per day;
* Has a positive test for antibody to human immunodeficiency virus (HIV-1 or -2) or hepatitis C virus;
* Has a positive test for hepatitis B surface antigen (HBsAg);
* Has at screening safety laboratory tests meeting one or more of the following criteria:
* hemoglobin < 10.5 g/dL
* white blood cell count < 4,000 cells/mm3
* absolute neutrophil count (ANC) < 1500/mm3
* platelet count < 100,000/mm3
* alanine transaminase (ALT; SGPT) > 1.5x ULN
* aspartate transaminase (AST; SGOT) > 1.5x ULN
* serum total bilirubin > 1.4x ULN
* serum creatinine > 1.3x ULN;
* Has a history of allogeneic organ transplant (including bone marrow or stem cells);
* Has, within the past 10 years, had evidence of or required treatment for cancer (except treated basal or squamous cell carcinoma of the skin or cured cervical carcinoma-in-situ);
* Has had within the past three months or is expected to have during the study period any of the following treatments:
* surgery requiring general anesthesia
* hematopoietic stimulating agents (e.g., erythropoietin, G-CSF, GM-CSF)
* another investigational drug;
* Has other significant medical disease (chronic or active within the past 6 months), including, but not limited to: cardiac disease (e.g., unstable angina, myocardial infarction, congestive heart failure, ventricular arrhythmia); uncontrolled seizure disorder; liver disease; chronic infection (e.g., tuberculosis); uncontrolled diabetes;
* Has any other condition that would, in the opinion of the Investigator, potentially compromise the safety or compliance of the patient or may preclude the patient's successful completion of the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Arbeit, MD, Study Director — Idera Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - Florida Center for Dermatology, P.A, Jacksonville, Florida
  - Atlanta Dermatology, Vein & Research Center, PC, Alpharetta, Georgia
  - Dermatologic Surgery Specialists, Inc., Macon, Georgia
  - Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - DermResearch PLLC, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Mass General Hospital Clinical Unit for Research Trials in Skin, Boston, Massachusetts
  - Derm Research Center of New York, Stony Brook, New York
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Clinical Partners, Inc, Johnston, Rhode Island
  - J & S Studies, College Station, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah, Dermatology, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 13 study centers in the Unites States (US).
Pre-assignment Details: 48 patients met inclusion/exclusion criteria; 4 were not randomized. The reasons for not randomizing these patients were: 2 patients withdrew consent, 1 whose calcium levels did not meet the criteria for randomization, and 1 for whom the study was closed prior to randomization
Period: Overall Study
Arm/Group | IMO-3100 at 0.16 mg/kg | IMO-3100 at 0.32 mg/kg | Placebo
Started | 15 | 14 | 15
Completed | 14 | 14 | 14
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | IMO-3100 at 0.16 mg/kg | IMO-3100 at 0.32 mg/kg | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 15 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13.76) | 41.9 (12.54) | 39.6 (13.15) | 39.6 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 11 | 28
  Male | 9 | 3 | 4 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 12 | 13 | 40
  Black | 0 | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Mean Epidermal Thickness at End-of-Treatment (EOT) Compared to Pre-treatment
Description: The change from pre-treatment baseline to End-of-Treatment (EOT) in the epidermal thickness of the index lesion
Time Frame: 8 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | IMO-3100 at 0.16 mg/kg | IMO-3100 at 0.32 mg/kg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Millimeters | -8.8 (85.9) | -48.5 (91.0) | 17.3 (102.8)

ADVERSE EVENTS:
Time Frame: AEs were collected from the first screening visit (Day -28) through the end of study visit (Day 60).
Description: An Adverse Event was defined as any untoward medical occurrence temporally associated with the use of a medical product in a subject. An AE could be a new occurrence or an existing process that increased significantly in intensity or frequency.
  * Unfavorable and unintended symptom reported by the subject;
  * Clinical sign detected by the Investigator;
  * Abnormal result from a laboratory study or other diagnostic procedure;
Arm/Group | IMO-3100 at 0.16 mg/kg | IMO-3100 at 0.32 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 6/15 | 8/14 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMO-3100 at 0.16 mg/kg (N=15) | IMO-3100 at 0.32 mg/kg (N=14) | Placebo (N=15)
Sclera hemorrhage (Eye disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Injection site discoloration (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Infected bites (Infections and infestations) | 0 | 1 | 0
Nasopharynghitis (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Anthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Albumin urine present (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hypoasthenia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes